CLINICAL TRIAL: NCT00607048
Title: A Phase 1 Study Of CP- 870,893 In Combination With Paclitaxel And Carboplatin In Patients With Metastatic Solid Tumors
Brief Title: Dose Finding Study Of CP-870,893, An Immune System Stimulating Antibody, In Combination With Paclitaxel And Carboplatin For Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5021004
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Paclitaxel; Carboplatin; selicrelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Schedule A (Other): Schedule A (CP-870,893 administration schedule)
  Interventions: Drug: Paclitaxel + Carboplatin + CP-870,893
- Schedule B (Other): Schedule B (CP-870,893 administration schedule)
  Interventions: Drug: Paclitaxel + Carboplatin + CP-870,893

INTERVENTIONS:
Drug: Paclitaxel + Carboplatin + CP-870,893 — Paclitaxel is administered intravenously on day 1 of a 21-day cycle at a dose of 175 mg/m^2. Carboplatin is administered intravenously on day 1 of a 21-day cycle at AUC 6. CP-870,893 is administered intravenously on DAY 3 of a 21-day cycle in escalating doses (0.1 mg/kg and 0.2 mg/kg)
  Arms: Schedule A
Drug: Paclitaxel + Carboplatin + CP-870,893 — Paclitaxel is administered intravenously on day 1 of a 21-day cycle at a dose of 175 mg/m^2. Carboplatin is administered intravenously on day 1 of a 21-day cycle at AUC 6. CP-870,893 is administered intravenously on DAY 8 of a 21-day cycle in escalating doses (0.1 mg/kg and 0.2 mg/kg)
  Arms: Schedule B

SUMMARY:
This is a dose-finding study; therefore, there is no hypothesis testing

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic solid tumors, for whom carboplatin and paclitaxel are appropriate;
* Patients >18 years of age;
* Good performance status;
* Adequate bone marrow and organ function

Exclusion Criteria:

* Previous treatment with any other compound that targets CD40
* Current or planned concurrent treatment with any anticancer agent;
* Patients who have received bone marrow transplant;
* History of autoimmune disorder
* History (within the previous year) of heart failure or heart attack
* Cancer-associated coagulation disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- [Derived] Vonderheide RH, Burg JM, Mick R, Trosko JA, Li D, Shaik MN, Tolcher AW, Hamid O. Phase I study of the CD40 agonist antibody CP-870,893 combined with carboplatin and paclitaxel in patients with advanced solid tumors. Oncoimmunology. 2013 Jan 1;2(1):e23033. doi: 10.4161/onci.23033. PMID 23483678

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 participants were screened, enrolled, and received at least 1 dose of study treatment in Schedule A. 18 participants were screened and enrolled in Schedule B; however, 2 participants discontinued before assignment to study treatment; 16 participants received at least 1 dose of study treatment in Schedule B.
Groups:
- Schedule A - CP-870893 0.1 mg/kg: Participants received fixed dose chemotherapy (carboplatin and paclitaxel) intravenously (IV) on Day 1 of every 21 day cycle.
  CP-870893 administered IV on Day 3 of every 21 day cycle with starting dose of 0.1 milligrams per kilogram (mg/kg) (0.1 mg/kg cohort).
- Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort): Participants received fixed dose chemotherapy (carboplatin and paclitaxel) IV on Day 1 of every 21 day cycle.
  If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.1 mg/kg cohort experienced a dose limiting toxicity in Cycle 1, subsequent participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 3 of every 21 day cycle (0.2 mg/kg escalation cohort).
- Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort): Participants received fixed dose chemotherapy (carboplatin and paclitaxel) IV on Day 1 of every 21 day cycle.
  If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.2 mg/kg cohort (escalation cohort) experienced a dose limiting toxicity in Cycle 1, 0.2 mg/kg was considered the maximum tolerated dose (MTD). Additional participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 3 of every 21 day cycle (0.2 mg/kg expansion cohort).
- Schedule B - CP-870893 0.1 mg/kg: Participants received fixed dose chemotherapy (carboplatin and paclitaxel) IV on Day 1 of every 21 day cycle.
  CP-870893 administered IV on Day 8 of every 21 day cycle with starting dose of 0.1 mg/kg (0.1 mg/kg cohort).
- Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort): Participants received fixed dose chemotherapy (carboplatin and paclitaxel) IV on Day 1 of every 21 day cycle.
  If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.1 mg/kg cohort experienced a dose limiting toxicity in Cycle 1, subsequent participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 8 of every 21 day cycle (0.2 mg/kg escalation cohort).
- Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort): Participants received fixed dose chemotherapy (carboplatin and paclitaxel) IV on Day 1 of every 21 day cycle.
  If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.2 mg/kg cohort (escalation cohort) experienced a dose limiting toxicity in Cycle 1, 0.2 mg/kg was considered the MTD. Additional participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 8 of every 21 day cycle (0.2 mg/kg expansion cohort).
Period: Overall Study
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Started | 3 | 6 | 7 | 3 | 6 | 7
Completed | 0 | 2 | 3 | 0 | 0 | 2
Not Completed | 3 | 4 | 4 | 3 | 6 | 5
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 4 | 0
Not completed — Global deterioration of health | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Objective disease progression - relapse | 1 | 2 | 4 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Other | 1 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Schedule A - CP-870893: Participants received fixed dose chemotherapy (carboplatin and paclitaxel) IV on Day 1 of every 21 day cycle.
  CP-870893 administered IV on Day 3 of every 21 day cycle with starting dose of 0.1 mg/kg (0.1 mg/kg cohort).
  If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.1 mg/kg cohort experienced a dose limiting toxicity in Cycle 1, subsequent participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 3 of every 21 day cycle (0.2 mg/kg escalation cohort).
  If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.2 mg/kg cohort (escalation cohort) experienced a dose limiting toxicity in Cycle 1, 0.2 mg/kg was considered the MTD. Additional participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 3 of every 21 day cycle (0.2 mg/kg expansion cohort).
- Schedule B - CP-870893: Participants received fixed dose chemotherapy (carboplatin and paclitaxel) IV on Day 1 of every 21 day cycle.
  CP-870893 administered IV on Day 8 of every 21 day cycle with starting dose of 0.1 mg/kg (0.1 mg/kg cohort).
  If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.1 mg/kg cohort experienced a dose limiting toxicity in Cycle 1, subsequent participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 8 of every 21 day cycle (0.2 mg/kg escalation cohort).
  If 0 out of 3 or <2 out of 6 participants in the CP-870893 0.2 mg/kg cohort (escalation cohort) experienced a dose limiting toxicity in Cycle 1, 0.2 mg/kg was considered the MTD. Additional participants were enrolled in the 0.2 mg/kg dose cohort and received CP-870893 0.2 mg/kg IV on Day 8 of every 21 day cycle (0.2 mg/kg expansion cohort).
- Total: Total of all reporting groups
Arm/Group | Schedule A - CP-870893 | Schedule B - CP-870893 | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (13.4) | 54.5 (12.7) | 56.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Cycle Dose Limiting Toxicities (DLTs)
Description: Any of the following during first cycle of treatment and attributable to CP-870893: Grade (Gr) 4 neutropenia (absolute neutrophil count [ANC] <500 cells/mm^3) for ≥7 days; Gr 3 or 4 febrile neutropenia (ANC <1000/mm^3, fever ≥38.5 degrees Celsius; platelets ≤25,000 cells/mm^3); ≥Gr 3 non-hematological adverse event despite optimal supportive care; ≥Gr 3 cytokine release syndrome or acute infusion reaction; failure to recover to Gr <1 toxicity after delaying next cycle by maximum of 2 weeks; Day 3 or 8 ANC <1000 cells/mm^3 or platelets <80000 cells/mm^3, or non-hematologic toxicity ≥Gr 2.
Time Frame: Schedule (Sch) A Cycle 1 / Day 3 or Schedule B Cycle 1 / Day 8 up to Cycle 1 / Day 21
Population: Safety population: all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 3 | 6 | 7 | 3 | 6 | 7
participants | 0 | 1 | 0 | 0 | 1 | 0

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: Mean of individual observed Cmax values measured as micrograms per milliliter (mcg/mL).
Time Frame: Schedule A Day 3 of each 21 Day Cycle, Schedule B Day 8 of each 21 Day Cycle: Pre-dose, 5 minutes after end of infusion, and 2, 6, and 24 hours (hrs) post-dose up to a maximum of 8 cycles (6 months)
Population: Pharmacokinetic data analysis set: all enrolled participants who started treatment and had baseline and sufficient on-study samples to provide interpretable results. N=number of participants who did not have pre-dose levels of CP-870893.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 3 | 6 | 7 | 2 | 6 | 7
mcg/mL | 0.97 (0.43) | 1.51 (0.60) | 1.36 (0.68) | 0.61 (NA) — Standard deviation not calculated for N <3. | 1.97 (0.99) | 1.06 (0.42)

3. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the serum concentration time-curve from time zero to the last measured concentration. AUClast was estimated using non-compartmental methods on the sequence of sample measurements. Mean of individual observed AUClast values measured as nanograms multiplied by micrograms per milliliter (ng*mcg/mL).
Time Frame: Schedule A Day 3 of each 21 Day Cycle, Schedule B Day 8 of each 21 Day Cycle: Pre-dose, 5 minutes after end of infusion, and 2, 6, and 24 hours post-dose up to a maximum of 8 cycles (6 months)
Population: Pharmacokinetic data analysis set; N=number of participants who did not have pre-dose levels of CP-870893.
Measure: Mean (Standard Deviation); unit: hr*mcg/mL
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 3 | 6 | 7 | 2 | 6 | 7
hr*mcg/mL | 3.37 (1.2) | 10.4 (9.3) | 7.5 (8.7) | 1.35 (NA) — Standard deviation not calculated for N <3. | 13.0 (10.3) | 5.71 (5.36)

4. Secondary Outcome: Tumor Response of Partial Response (PR) and Complete Response CR) According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Number of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as the disappearance of all target and nontarget lesions. PR was defined as a ≥30% decrease in the sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD.
Time Frame: Schedule A and Schedule B: Baseline and Day 21 of every even numbered cycle up to a maximum of 8 cycles (6 months)
Population: All response-evaluable population: included all participants who had measurable disease, a baseline tumor assessment and who started treatment were considered evaluable for analysis of tumor response.
Measure: Number; unit: participants
Arm/Group | Schedule A - CP-870893 | Schedule B - CP-870893
Number analyzed (Participants) | 16 | 16
participants
  Complete response | 0 | 0
  Partial response | 2 | 3

5. Secondary Outcome: Change in Cytokine Concentrations of Interleukin 6 (IL 6): Pre-dose Concentration (CYTO0), Maximum Post-dose Concentration (CYTOMAX)
Description: Concentrations reported as the mean of the pre-dose values and the mean of the maximum post-dose values to show change. An increase in values indicates greater cytokine release from cells targeted by the antibody and may be associated with an infusion reaction.
Time Frame: Schedule A Cycle 1 / Day 3 and Schedule B Cycle 1 / Day 8: predose, end of infusion, 1 , 2, 4, 6, 24, and 48 hours postdose
Population: Pharmacokinetic data analysis set.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 3 | 6 | 7 | 3 | 6 | 7
picograms per milliliter (pg/mL)
  CYTO0 | 10.57 (5.8106) | 12.10 (9.5896) | 14.52 (14.674) | 3.547 (0.7390) | 41.34 (72.595) | 8.040 (6.6632)
  CYTOMAX | 120.67 (92.5545) | 275.48 (427.617) | 371.22 (379.799) | 113.45 (42.1629) | 339.00 (185.140) | 679.40 (856.849)

6. Secondary Outcome: Change in Cytokine Concentrations of Tumor Necrosis Factor Alpha (TNF Alpha): CYTO0, CYTOMAX
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Pharmacokinetic data analysis set. CYTO0 values = the lower limit of quantitation (LLOQ).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 3 | 6 | 7 | 3 | 6 | 7
pg/mL
  CYTO0 | 15.60 (0.0000) | 15.60 (0.0000) | 15.60 (0.0000) | 15.60 (0.0000) | 15.60 (0.0000) | 15.60 (0.0000)
  CYTOMAX | 155.73 (151.527) | 108.90 (148.896) | 113.11 (75.4270) | 212.73 (166.857) | 161.90 (196.651) | 675.34 (1263.56)

7. Secondary Outcome: Change in Bone Marrow Derived Cells (B Cell) Surface Markers: CD19 Pre-dose Percentage (PD0), Maximum Post-dose Percentage (PDmax)
Description: Assess activity of B cells (involved in production of antibodies) in presence of CP-870893. Clusters of differentiation (CD) are specific types of proteins on cell surface. CD19 is a B cell antigen receptor and is used to quantitate changes in proportion of B cells in peripheral blood as a consequence of therapy. Higher numbers may indicate a greater presence of CD19 on cell surface with increased potential for antigen response. Percentage of cells reported as the mean of the pre-dose values and the mean of the maximum post-dose values to show change.
Time Frame: Schedule A Cycle 1 / Day 3 and Schedule B Cycle 1 / Day 8: predose, 6, 24, and 48 hours postdose
Population: Biomarker data analysis set: All enrolled participants who started treatment and who had baseline and sufficient on-study samples to provide interpretable results. N=Number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 2 | 6 | 7 | 3 | 6 | 7
percentage of cells
  PD0 | 5.81 (1.4284) | 9.12 (5.2037) | 11.3257 (6.1987) | 13.5233 (13.8885) | 9.42 (5.1037) | 6.5514 (3.3797)
  PDMAX | 4.99 (0.9758) | 7.3017 (5.1317) | 9.4614 (5.0745) | 6.7133 (3.8467) | 7.7783 (4.4316) | 4.6786 (2.9114)

8. Secondary Outcome: Change in Bone Marrow Derived Cells (B Cell) Surface Markers: CD40 PD0, PDmax
Description: Assess activity of B cells in the presence of CP-870893. CD40 is a costimulatory protein and is a target for CP-870893. Measurement of CD40 on white blood cells provides a measure of target modulation by CP-870893. Higher numbers may indicate potential for increased activation of antigen presenting cells. Percentage of cells reported as the mean of the pre-dose values and the mean of the maximum post-dose values to show change.
Time Frame: Schedule A Cycle 1 / Day 3 and Schedule B Cycle 1 / Day 8: predose, 6, 24, and 48 hours postdose
Population: Biomarker data analysis set; N=Number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 2 | 6 | 7 | 3 | 6 | 7
percentage of cells
  PD0 | 99.265 (0.7566) | 99.8267 (0.2447) | 99.0043 (1.4442) | 99.9833 (0.0289) | 99.6533 (0.4772) | 88.07 (28.0802)
  PDMAX | 6.615 (8.2237) | 11.7883 (17.8460) | 13.6929 (27.7995) | 0.65 (0.6497) | 18.9517 (38.0439) | 12.6514 (26.8913)

9. Secondary Outcome: Change in Bone Marrow Derived Cells (B Cell) Surface Markers: CD23 PD0, PDmax
Description: Assess activity of B cells in the presence of CP-870893. CD23 is a low-affinity receptor that has a role in transportation in antibody feedback regulation. Agents that engage CD40 have been reported to increase CD23 expression; increased CD23 expression may, therefore, serve as a marker for CD40 binding by CP-870893. Higher numbers may indicate a potential for increased antibody response. Percentage of cells reported as the mean of the pre-dose values and the mean of the maximum post-dose values to show change.
Time Frame: Schedule A Cycle 1 / Day 3 and Schedule B Cycle 1 / Day 8: predose, 6, 24, and 48 hours postdose
Population: Biomarker data analysis set; N=Number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 2 | 6 | 7 | 3 | 6 | 7
percentage of cells
  PD0 | 71.155 (16.3554) | 86.2267 (8.7526) | 80.4843 (14.5377) | 90.2333 (5.0997) | 85.26 (5.2701) | 83.0943 (8.7534)
  PDMAX | 22.155 (14.2765) | 36.735 (30.9453) | 20.0857 (8.1089) | 7.58 (4.8650) | 22.3183 (17.2221) | 33.3057 (24.0570)

10. Secondary Outcome: Change in Bone Marrow Derived Cells (B Cell) Surface Markers: CD54 PD0, PDmax
Description: Assess activity of B cells in presence of CP-870893. CD54 is an intercellular adhesion molecule. When activated, leukocytes bind to endothelial cells via CD54 and then transmigrate into tissues. Agents that engage CD40 have been reported to increase CD54 expression; increased CD54 expression may, therefore, serve as a marker for CD40 binding by CP-870893. Higher numbers may indicate potential for increased immune response. Percentage of cells reported as the mean of the pre-dose values and the mean of the maximum post-dose values to show change.
Time Frame: Schedule A Cycle 1 / Day 3 and Schedule B Cycle 1 / Day 8: predose, 6, 24, and 48 hours postdose
Population: Biomarker data analysis set; N=Number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 2 | 6 | 7 | 3 | 6 | 7
percentage of cells
  PD0 | 95.735 (5.8902) | 94.7667 (9.0938) | 97.9486 (0.8686) | 99.6367 (0.3465) | 96.4867 (3.7710) | 94.5571 (2.9589)
  PDMAX | 28.505 (32.0532) | 25.85 (25.9993) | 23.5229 (15.4014) | 1.7 (1.5156) | 33.2017 (33.3072) | 21.1886 (33.3022)

11. Secondary Outcome: Change in Bone Marrow Derived Cells (B Cell) Surface Markers: CD86 PD0, PDmax
Description: Assess activity of B cells in presence of CP-870893. CD86 is a protein expressed on antigen-presenting cells and provides co-stimulatory signals for T cell (role in cell-modulated immunity) activation. Agents that engage CD40 have been reported to increase CD86 expression; increased CD86 expression may, therefore, serve as a marker for CD40 binding by CP-870893. Higher numbers may indicate potential for increased immune response. Percentage of cells reported as the mean of the pre-dose values and the mean of the maximum post-dose values to show change.
Time Frame: Schedule A Cycle 1 / Day 3 and Schedule B Cycle 1 / Day 8: predose, 6, 24, and 48 hours postdose
Population: Biomarker data analysis set; N=Number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 2 | 6 | 7 | 3 | 6 | 7
percentage of cells
  PD0 | 3.91 (0.4384) | 5.8167 (3.4037) | 18.7629 (8.2298) | 5.5367 (4.4152) | 9.23 (5.1565) | 16.7186 (5.4602)
  PDMAX | 12.795 (3.0618) | 26.275 (23.1242) | 11.9443 (10.3140) | 18.04 (19.9811) | 28.0917 (16.5569) | 34.3943 (18.5593)

12. Secondary Outcome: Change in Bone Marrow Derived Cells (B Cell) Surface Markers: Human Leukocyte Antigen (HLA-DR) PD0, PDmax
Description: Assess activity of B cells in presence of CP-870893. HLA-DR is a component of the Major Histocompatibility Complex in humans and presents antigens for recognition by the immune system. Agents that engage CD40 have been reported to increase HLA-DR expression; increased HLA-DR expression may serve as a marker for CD40 binding by CP-870893. Positive values may indicate greater presence of cells associated with potential for antibody production. Percentage of cells reported as the mean of the pre-dose values and the mean of the maximum post-dose values to show change.
Time Frame: Schedule A Cycle 1 / Day 3 and Schedule B Cycle 1 / Day 8: predose, 6, 24, and 48 hours postdose
Population: Biomarker data analysis set; N=Number of participants contributing to the mean.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 2 | 6 | 7 | 3 | 6 | 7
percentage of cells
  PD0 | 98.24 (2.1355) | 98.325 (1.9341) | 99.0986 (0.4929) | 99.7833 (0.2021) | 97.4 (3.4616) | 98.5643 (1.8466)
  PDMAX | 33.88 (38.3818) | 27.4983 (24.3301) | 21.7857 (12.1245) | 2.7833 (2.5010) | 15.1783 (20.5400) | 27.0986 (33.2939)

13. Secondary Outcome: Total and Neutralizing Human Antihuman Antibody (HAHA) Titer
Description: HAHA assessed as an indicator of immunogenicity to CP-870893.
Time Frame: Schedule A Day 3 of each 21 Day Cycle, Schedule B Day 8 of each 21 Day Cycle: Pre-dose up to a maximum of 8 cycles (6 months)
Population: Data was not summarized as Human antihuman responses to CP-870893 were all below the limit of quantitation (endpoint titer of 4.32).
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are reported from the time of the first dose of study treatment up to 43 days after last dose of study treatment.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Schedule A - CP-870893 0.1 mg/kg | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) | Schedule B - CP-870893 0.1 mg/kg | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort)
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/6 | 2/7 | 0/3 | 3/6 | 2/7
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 7/7 | 3/3 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A - CP-870893 0.1 mg/kg (N=3) | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) (N=6) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) (N=7) | Schedule B - CP-870893 0.1 mg/kg (N=3) | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) (N=6) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort) (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Optic nerve infarction (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A - CP-870893 0.1 mg/kg (N=3) | Schedule A - CP-870893 0.2 mg/kg (Escalation Cohort) (N=6) | Schedule A - CP-870893 0.2 mg/kg (Expansion Cohort) (N=7) | Schedule B - CP-870893 0.1 mg/kg (N=3) | Schedule B - CP-870893 0.2 mg/kg (Escalation Cohort) (N=6) | Schedule B - CP-870893 0.2 mg/kg (Expansion Cohort) (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 3 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 2 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 2 | 4
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2 | 3
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 1 | 1 | 1 | 2
Fatigue (General disorders) | 3 | 5 | 6 | 2 | 4 | 6
Infusion site extravasation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mucosal haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 0 | 3 | 2
Cytokine release syndrome (Immune system disorders) | 2 | 3 | 2 | 1 | 3 | 3
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 2 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0 | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 3
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 4 | 0 | 2 | 6
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 6 | 2 | 1 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.